CLINICAL TRIAL: NCT04277429
Title: The Influence of hearT Failure With Preserved Ejection Fraction on 2year Mortality of Patients With cHronic obstructivE pulmonaRy disEaSE- THERESE Study
Brief Title: HFpEF and 2-year Mortality of COPD Patients
Acronym: THERESE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Milan Sova, Principal Investigator, Department of Respiratory Medicine, University Hospital Olomouc
Other Study IDs: THERESE
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal cardiac function: Normal cardiac function
  Interventions: Diagnostic Test: Cardiac function assessment
- Heart failure with reduced ejection fraction: Heart failure with reduced ejection fraction
  Interventions: Diagnostic Test: Cardiac function assessment
- Heart failure with preserved ejection fraction: Heart failure with preserved ejection fraction
  Interventions: Diagnostic Test: Cardiac function assessment

INTERVENTIONS:
Diagnostic Test: Cardiac function assessment — Echocardiography, cardiac enzymes analysis

SUMMARY:
This study was designed to assess potential relationship between heart failure with preserved ejection fraction and 2- year mortality of patients with chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

Exacerbation of chronic obstructive pulmonary disease requiring hospitalization

Age 40 - 80 years

Performance status 0-1 according to Eastern Cooperative Oncology Group (ECOG)

Long acting beta agonist (LABA)/ long acting antimuscarinic (LAMA) bronchodilator treatment

Exclusion Criteria:

Presence of major heart valve dysfunction

Documented noncompliance with treatment

Presence of active malignancy

Body mass index > 40

Interstitial lung disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 year
  Mortality of patients

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sova, Ph.D., Principal Investigator — Department of Respiratory Medicine
Locations (2):
- Czechia (2):
  - Frydek Mistek Hospital, Frýdek-Místek
  - University Hospital Olomou, Olomouc